CLINICAL TRIAL: NCT06876636
Title: Prospective, Open-Label, Single-Arm Clinical Study of Zoledronic Acid Combined With Neoadjuvant Chemotherapy (EC-T) in Patients With Early-Stage and Locally Advanced Triple-Negative Breast Cancer
Brief Title: Zoledronic Acid Combined With EC-T for Triple-Negative Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252004-C-1
Record Dates: First submitted 2025-02-26; First posted 2025-03-14 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Metastatic
Keywords: Zoledronic Acid; Neoadjuvant Chemotherapy
MeSH Terms: interventions — Neoadjuvant Therapy; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zoledronic Acid (Experimental): Zoledronic acid 4 mg on Day 1 every 3 weeks (q3w) plus liposomal doxorubicin 35 mg/m² on Day 1 q3w plus cyclophosphamide 600 mg/m² on Day 1 q3w, for four cycles. Concurrent immunotherapy is permitted: pembrolizumab 200 mg on Day 1 q3w or toripalimab 240 mg on Day 1 q3w.
  Thereafter, zoledronic acid 4 mg on Day 1 q3w plus nab-paclitaxel 260 mg/m² on Day 1 q3w for another four cycles. If immunotherapy was given during the first four cycles, it may be continued for the latter four cycles.
  A total of eight chemotherapy cycles are planned, with allowance for multiple drug interruptions due to adverse events.
  Interventions: Drug: Zoledronic Acid Combined with Neoadjuvant Chemotherapy (EC-T)

INTERVENTIONS:
Drug: Zoledronic Acid Combined with Neoadjuvant Chemotherapy (EC-T) — zoledronic acid + liposomal doxorubicin + cyclophosphamide followed by zoledronic acid + nab-paclitaxel Concurrent immunotherapy is permitted: pembrolizumab or toripalimab
  Other Names: Zoledronic Acid

SUMMARY:
Exploring the efficacy and safety of zoledronic acid combined with neoadjuvant chemotherapy (EC-T) in neoadjuvant treatment for early-stage or locally advanced triple-negative breast cancer, the trial protocol of zoledronic acid + liposomal doxorubicin + cyclophosphamide followed by zoledronic acid + nab-paclitaxel will provide a new effective therapeutic strategy for neoadjuvant treatment of triple-negative breast cancer patients and offer a novel treatment approach for triple-negative breast cancer.

DETAILED DESCRIPTION:
This study is a prospective, open-label, single-arm clinical trial, planning to enroll 99 treatment-naïve patients with early-stage or locally advanced triple-negative breast cancer (clinical stage IIA-IIIC). The neoadjuvant treatment regimen consists of four cycles of chemotherapy with zoledronic acid + liposomal doxorubicin + cyclophosphamide, followed by four cycles of chemotherapy with zoledronic acid + nab-paclitaxel. The study aims to explore the efficacy and safety of zoledronic acid combined with neoadjuvant chemotherapy (EC-T) in the neoadjuvant treatment of early-stage or locally advanced triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years and ≤75 years who have not received prior treatment;
2. ECOG score of 0 to 1;
3. Her-2 (0), Her-2 (1+), Her-2 (2+) must test negative by ISH (in situ hybridization).
4. Hormone receptor status: ER (Estrogen Receptor) <1%, PR (Progesterone Receptor) <1%;
5. The functional levels of major organs must meet the following requirements (no blood transfusion within 2 weeks prior to screening, no use of white blood cell or platelet-raising drugs):
6. Complete blood count： Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥90×10^9/L; Hemoglobin (Hb) ≥90 g/L;
7. Blood chemistry Total bilirubin (TBIL) ≤ upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5×ULN; Alkaline phosphatase ≤2.5×ULN; Blood urea nitrogen (BUN) and creatinine (Cr) ≤1.5×ULN;
8. Echocardiogram Left ventricular ejection fraction (LVEF) ≥55%; 9、12-lead ECG QTc interval corrected by Fridericia's method (QTcF) <470 msec.

10、For premenopausal or surgically unsterilized female patients: agree to abstain from sexual intercourse or use effective contraceptive methods during the treatment period and for at least 7 months after the last administration of study treatment.

11、Voluntarily participate in this study, sign the informed consent form, have good compliance, and are willing to cooperate with follow-up visits

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer;
2. Inflammatory breast cancer;
3. A history of receiving anti-cancer treatment or radiotherapy for any malignant tumor, excluding curative treatments for in situ cervical cancer, basal cell carcinoma, or squamous cell carcinoma, etc.;
4. Concurrently participating in other clinical trials involving anti-cancer therapies, including endocrine therapy, bisphosphonate therapy, or immunotherapy;
5. Having undergone significant non-breast cancer related surgical procedures within 4 weeks prior to enrollment, or not having fully recovered from such procedures;
6. Severe cardiac disease or conditions, including but not limited to the following:

   * A confirmed history of heart failure or systolic dysfunction (LVEF <50%);
   * High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate >100 bpm, significant ventricular arrhythmias (e.g., ventricular tachycardia), or higher-grade atrioventricular block (i.e., Mobitz Type II second-degree atrioventricular block or third-degree atrioventricular block);
   * Angina requiring anti-anginal medication;
   * Clinically significant valvular heart disease;
   * ECG showing transmural myocardial infarction;
   * Poorly controlled hypertension (systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg);
7. Inability to swallow, intestinal obstruction, or other factors affecting drug intake and absorption;
8. Known history of allergies to the components of the study medication: a history of immunodeficiency, including positive HIV tests, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
9. Pregnant or nursing women, women of childbearing potential with a positive baseline pregnancy test, or women of reproductive age who are unwilling to use effective contraceptive measures throughout the trial period and for 7 months after the last administration of study medication;
10. Having severe concomitant diseases or other conditions that would interfere with planned treatment, or any other circumstances deemed by the investigator to make the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate | up to 6 months
  pCR is defined as the absence of invasive tumor cells in the breast and axillary lymph nodes after primary tumor resection (ypT0/is ypN0) as assessed microscopically.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 6 months
  The proportion of patients evaluated as having a Complete Response (CR) or Partial Response (PR) according to RECIST version 1.1.
Clinical Benefit Rate (CBR) | up to 6 months
  The proportion of patients evaluated as having a CR, PR, or Stable Disease (SD) lasting at least 6 months according to RECIST version 1.1.
Disease-Free Survival (DFS) | up to 6 years
  The time from enrollment to the first occurrence of recurrent disease, which includes ipsilateral or contralateral recurrence of breast cancer, local or regional recurrence, distant metastasis, and death from any cause.
Overall Survival (OS) | up to 6 years
  The time from enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No